CLINICAL TRIAL: NCT06665373
Title: A Pilot Study to Investigate the Effects of Combining a Modified Atkins Diet With a Physical Fitness Regimen in Patients Diagnosed With Malignant Glioma
Brief Title: Fitness and Nutrition in Glioma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-00654
Record Dates: First submitted 2024-10-29; First posted 2024-10-30 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Malignant Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients Diagnosed with Malignant Glioma (Experimental): Patients will participate in a 15-week program consisting of two weekly supervised exercise sessions combined with an individualized home exercise program and a modified Atkins diet.
  Interventions: Behavioral: Modified Atkins Diet; Behavioral: Fitness Program

INTERVENTIONS:
Behavioral: Modified Atkins Diet — The Atkins diet is a low-carb eating plan that focuses on balancing protein, fat, and carbohydrates.
Behavioral: Fitness Program — 12 weeks of two weekly supervised exercise sessions combined with an individualized home exercise program based on physical capabilities and available equipment.

SUMMARY:
This is a pilot study assessing the effects of combining a modified Atkins diet with a physical fitness regimen in patients with malignant glioma. A sample size of 15 participants will be enrolled in a 15-week program consisting of two weekly supervised exercise sessions combined with an individualized home exercise program and a modified Atkins diet.

ELIGIBILITY:
Inclusion Criteria:

* Tissue confirmed diagnosis of high-grade glioma (World Health Organization grade III or IV)
* Karnofsky Performance Status (KPS) ≥ 70%
* Willing to follow the study intervention and follow-up
* Able to give full informed consent

Exclusion Criteria:

* Currently undergoing initial concurrent radiation/chemotherapy
* Severe medical co-morbidities
* Any medical condition which prohibits moderate to vigorous physical activity (60-85% HRmax)
* Any medical condition which prohibits a restrictive diet
* Neurological deficit preventing participation in moderate to vigorous physical activity
* Severe psychiatric illness

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change in Short Form (SF)-36 Version 2 Score | Baseline, Week 12
  The SF-36
Number of Participants who Complete Full 12-Week Program | Week 12

SECONDARY OUTCOMES:
Change in Blood Ketone Levels | Baseline, Week 12
Change in Resting Heart Rate | Baseline, Week 12
Change in 400-meter Walk Time | Baseline, Week 12
  Time to complete 400-meter-long distance corridor walk.
Change in 1 Repetition Maximum (1RM) - Chest Press | Baseline, Week 12
  The 1RM for chest press is the maximum weight an individual can perform for a chest press for one repetition.
Change in 1 Repetition Maximum (1RM) - Leg Press | Baseline, Week 12
  The 1RM for chest press is the maximum weight an individual can perform for a leg press for one repetition.
Change in Satisfaction With Life Scale (SWLS) Score | Baseline, Week 12
  5-item assessment of satisfaction with life. Each item is rated on a 7-point Likert scale. The total score is the sum of responses and ranges from 5-35; higher scores indicate greater satisfaction.
Change in Hospital Anxiety And Depression Scale (HADS) - Anxiety Subscale Score | Baseline, Week 12
  The HADS is a self-report rating scale of 14 items on a 4-point Likert scale (range 0-3). It is designed to measure anxiety and depression (7 items for each subscale). The total score for the Anxiety subscale is the sum of the respective seven items. The total score ranges from 0-21; higher scores indicate greater anxiety.
Change in Hospital Anxiety And Depression Scale (HADS) Score | Baseline, Week 12
  The HADS is a self-report rating scale of 14 items on a 4-point Likert scale (range 0-3). It is designed to measure anxiety and depression (7 items for each subscale). The total score is the sum of the items; the total score ranges from 0-42; higher scores indicate greater anxiety and depression.
Change in Fatigue Severity Scale (FSS) Score | Baseline, Week 12
  The Fatigue Severity Scale (FSS) is a 9-item questionnaire that measures the severity of fatigue and how it affects a person's lifestyle and activities. Items are rated on a 7-point Likert scale. The total score is the sum of responses and ranges from 9 to 63. A higher score indicates greater fatigue severity.

CONTACTS AND LOCATIONS:
Overall Officials: Lee Tessler, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Deidentified data will not be shared with other researchers